CLINICAL TRIAL: NCT01939509
Title: Comparison of the Hemodynamic Changes in Patients Under Treatment With Bisoprolol Versus Atenolol
Brief Title: Hemodynamic Changes of Patients Receiving Atenolol/Bisoprolol
Acronym: CHAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Lucas Aparicio, MD, Hospital Italiano de Buenos Aires
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1445
Record Dates: First submitted 2012-02-01; First posted 2013-09-11 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension; Metabolic Syndrome
MeSH Terms: conditions — Hypertension; Metabolic Syndrome | interventions — Atenolol; Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atenolol-Bisoprolol (Experimental)
  Interventions: Drug: Atenolol; Drug: Bisoprolol

INTERVENTIONS:
Drug: Atenolol — Crossover (atenolol 25-50 mg, bisoprolol 2.5-5 mg)
Drug: Bisoprolol

SUMMARY:
At hemodynamic level, the greater affinity of bisoprolol by the beta 1 receptor in theory could improve the peripheral arterial perfusion and could have a greater antihypertensive effect. At the same time, this could carry objectifiable improvements in the vascular tree, such as the level of arterial stiffness.

This study attempts to mark the hemodynamic differences in the same individual with hypertension and metabolic syndrome who will be exposed to both drugs at different moments. Parameters will be objectified with impedance cardiography, pulse wave velocity and central blood pressure assessment before and after taking each one of the drugs. The results will be compared to the baseline data and between themselves.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension
* Metabolic syndrome

Exclusion Criteria:

* Severe hypertension >180/110
* Secondary hypertension
* Contraindication for betablockers
* Prior treatment with betablockers (up to one month before inclusion)
* History of neoplastic disease
* Patients that do not sign informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
central blood pressure | two months

SECONDARY OUTCOMES:
peripheral resistance | two months
cardiac index | two months
pulse wave velocity | two months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel D Waisman, MD, Study Director — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina